CLINICAL TRIAL: NCT05975008
Title: Pilot Testing a Virtual Mindfulness-Based Intervention Aimed at Improving Reintegrating Veterans' Health Outcomes
Brief Title: Pilot Testing a Virtual Mindfulness-Based Intervention to Improve Veterans' Health
Acronym: RECLAIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PPO 22-150
Record Dates: First submitted 2023-07-25; First posted 2023-08-03 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Depression
Keywords: mindfulness; mental health; community reintegration
MeSH Terms: conditions — Depression; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This is a pilot randomized controlled trial. Intervention arm participants will participate in the 8-week intervention. Control group participants will receive psychoeducation materials that the intervention group will also receive.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RECLAIM intervention (Experimental): Eight sessions of a brief mindfulness-based intervention that meets weekly in a virtual setting.
  Interventions: Behavioral: RECLAIM - Reconnecting to Civilian Life using Activities that Improve Mindfulness
- Psychoeducation materials only (No Intervention): The investigators will use a psychoeducation-only control group. They will only receive psychoeducational materials (e.g., suggested readings, podcasts, blogs). These are the same materials that the intervention arm participants will receive.

INTERVENTIONS:
Behavioral: RECLAIM - Reconnecting to Civilian Life using Activities that Improve Mindfulness — Brief virtual mindfulness-based intervention
  Arms: RECLAIM intervention

SUMMARY:
The purpose of this study is to test a mindfulness-based intervention to reduce depressive symptoms and improve Veterans' community reintegration.

DETAILED DESCRIPTION:
The overarching goal of the proposed project is to use mindfulness practices to reduce depression and improve community reintegration among post-9/11 Veterans. This proposal focuses on the REconnecting to Civilian Life using Activities that Improve Mindfulness (RECLAIM) intervention. RECLAIM is a virtual multi-component, mindfulness-based intervention developed by the study team in collaboration with VA clinicians, post-9/11 Veterans, and stakeholders and guided by the VA Whole Health framework. The proposed project builds on preliminary pilot work and a Small Award Initiative for Impact (SWIFT) pilot project funded by the VA HSR&D Center of Innovation. In the SWIFT pilot, the investigators refined the RECLAIM content and tested the feasibility of virtual delivery with a small sample (N=18) using a single arm pre/post-test design. The proposed pilot project builds on preliminary work by (1) testing the refined intervention in a randomized controlled design to assess feasibility of recruitment for a randomized trial, (2) randomization, (3) retention in both study arms, and (4) intervention acceptability. Findings from the proposed project will support a HSR&D Investigator Initiated Research Merit award application that will assess the effectiveness of RECLAIM while simultaneously planning for implementation in a Hybrid Type I trial. The following are the specific aims for this pilot project.

Aim 1: Conduct a randomized controlled pilot study to assess feasibility of the RECLAIM intervention. The investigators will conduct a two-arm randomized pilot study. Veterans (N=48) will be randomized to either the intervention arm (i.e., virtually delivered RECLAIM) or a control arm (i.e., psychoeducation materials). The investigators will assess intervention feasibility, including recruitment, randomization, administration and completion of outcome assessments, treatment engagement, and retention in both the intervention and control study arms.

Aim 2: Conduct qualitative interviews to assess acceptability of RECLAIM. A purposefully sampled subgroup (i.e., based on attendance) of RECLAIM participants (i.e., Veterans from the intervention arm; N=16) will engage in a qualitative interview to explore experiences in RECLAIM, including perceived strengths and suggestions for future improvements.

Aim 3: Refine and finalize the RECLAIM intervention. As findings emerge from the Aim 1 pilot test and Aim 2 interviews with Veteran participants, the investigators will iteratively update the RECLAIM protocol manual and testing procedures (i.e., randomization, control group materials). The investigators will consult with the Patient Advisory Council of the Indianapolis VAMC to gather Veteran feedback on the revised RECLAIM protocol manual, as well as partners (e.g., Patient Centered Care and Cultural Transformation). These actions will help refine the study methods, design, and intervention in anticipation of a larger trial.

ELIGIBILITY:
Inclusion Criteria:

Veteran participants must:

* be between 18-44 years old
* have served (a) active duty and/or (b) in the National Guard/Reserves, after October 2001 (can still be in the National Guard or Reservist)
* be enrolled in VHA care
* endorse at least "some" difficulty adjusting to civilian life to be eligible for participation. Difficulty adjusting to civilian life (i.e., reintegration challenges) will be assessed using the Military to Civilian Questionnaire (M2C-Q). For this study, "some" difficulty will be defined as a mean M2C-Q score of 2; the M2C-Q developers established a score of 2 as indicative of "some" reintegration difficulty and, as such, this is the score the investigators will use in the current study.
* endorse at least a moderate level of depression. The investigators will use the Patient Health Questionnaire (PHQ-9). to assess the presence and severity of depressive symptoms among potential Veteran participants. Moderate depression is defined as a score of 10-14 on the PHQ-9. This strategy for eligibility criteria optimally positions us to target Veterans who will likely benefit most from RECLAIM and to detect intervention effects in a future fully-powered follow-up trial.

Exclusion Criteria:

* Veterans will not be immediately excluded from participation in the study; the study team will consult with the Roudebush Suicide Prevention Team and/or the Veterans' care provider to determine whether continued study participation is appropriate.

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah A Shue, PhD MS BA, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (1):
- Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The investigators requested a list of Veterans and their contact information based on the study inclusion criteria via CDW. The research assistant mailed a recruitment brochure and letter to eligible Veterans. Study staff contacted eligible Veteran participants by phone and/or email to recruit them for the study. Veterans who enrolled were emailed using VA compliant methods. Word-of-mouth and snowballing techniques were also used to identify eligible Veteran participants.
Pre-assignment Details: Some participants were lost to follow-up (i.e., could not be contacted after enrolling in the study) or withdrew due to scheduling conflicts.
Groups:
- RECLAIM/Intervention: Veteran participants randomized to the intervention group. Eight sessions of a brief mindfulness-based intervention that meets weekly in a virtual setting.
- Psychoeducation Materials Only/Control Group: The investigators will use a psychoeducation-only control group. They will only receive psychoeducational materials (e.g., suggested readings, podcasts, blogs). These are the same materials that the intervention arm participants will receive.
Period: Overall Study
Arm/Group | RECLAIM/Intervention | Psychoeducation Materials Only/Control Group
Started | 18 | 18
Completed | 8 | 7
Not Completed | 10 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RECLAIM/Intervention | Psychoeducation Materials Only/Control Group | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.1 (7.3) | 30 (6) | 30.5 (6.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 11 | 14 | 25
  Gender: Female | 6 | 4 | 10
  Gender: Not disclosed | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 17 | 13 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 12 | 14 | 26
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 0 | 1 | 1
Military to Civilian Questionnaire [Mean (Standard Deviation); unit: score on a scale] — The Military to Civilian Questionnaire (M2CQ) is a 16-item self-report tool assessing difficulties in areas like social relationships, work/school, self-care, and community engagement over the past 30 days using a 0-4 Likert scale (no to extreme difficulty) to gauge post-deployment reintegration. Scores can range from 0-64. Higher scores indicate greater reintegration difficulty.
  score on a scale | 36.3 (12.7) | 33.3 (7.5) | 34.9 (10.4)
Patient Health Questionnaire [Mean (Standard Deviation); unit: score on a scale] — The Patient Health Questionnaire (PHQ-9) is a set of self-report questions to screen, diagnose, monitor, and measure the severity of depression symptoms. The PHQ-9 consists of 9 questions, each focusing on depressive symptoms over the past 2 weeks. Scores can range from 0-27 and higher scores indicate greater depression severity.
  score on a scale | 15.9 (5.8) | 13.6 (3.6) | 14.3 (4.8)
Generalized Anxiety Disorder Scale [Mean (Standard Deviation); unit: score on a scale] — The Generalized Anxiety Disorder Scale (GAD-7) is a brief, self-administered screening tool used to measure the presence and severity of anxiety symptoms. It consists of 7 questions and has a total score range from 0-21 and higher scores indicate greater frequency of anxiety symptoms.
  score on a scale | 12.6 (4.4) | 14.1 (5.2) | 13.5 (4.2)
Pain, Enjoyment, General Activity [Mean (Standard Deviation); unit: score on a scale] — The Pain, Enjoyment, and General Activity (PEG) scale is a three-item assessment tool used to monitor chronic pain over time. Each item uses a numerical rating scale from 0 to 10. The scores on each of the 3 items (pain levels on average, pain interference with enjoyment, and pain interference with general activity) are summed and averaged to provide a score that will range from 0-10. Lower scores indicate minimal pain impact.
  score on a scale | 4.4 (2.7) | 5.1 (2.1) | 4.7 (2.4)
Five Facet Mindfulness Questionnaire [Mean (Standard Deviation); unit: score on a scale] — The Five Facet Mindfulness Questionnaire (FFMQ-15) is a self-report scale that measures an individual's dispositional mindfulness across 5 distinct facets. Responses are made on a 5-point Likert scale, are totaled, and higher scores indicate greater mindfulness. The minimum possible score for each of the mindfulness facets is 3 and the maximum possible score is 15.
  score on a scale
    Facet of Mindfulness: Observing | 11 (4.1) | 9.0 (3.5) | 10.1 (3.9)
    Facet of Mindfulness: Describing | 9.5 (2.9) | 8.4 (2.2) | 9 (2.6)
    Facet of Mindfulness: Awareness | 10.5 (2) | 7.7 (2.6) | 9.2 (2.6)
    Facet of Mindfulness: Non-judging | 9 (3.7) | 9.3 (1.3) | 9.1 (2.7)
    Facet of Mindfulness: Non-reacting | 8.1 (2.5) | 9.1 (3.6) | 8.6 (3)

OUTCOME MEASURES:

1. Primary Outcome: Military to Civilian Questionnaire
Description: The Military to Civilian Questionnaire (M2C-Q) is an empirically validated self-report scale that measures general difficulty in readjusting to civilian life by assessing important indicators of reintegration challenges over the past 30 days including social/health behaviors, specifically interpersonal relationships; productivity at school, work, or home; community participation; self-care; leisure; and perceived meaning in life. Scores can range from 0-64. Higher scores indicate greater reintegration difficulty.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RECLAIM/Intervention | Psychoeducation Materials Only/Control Group
Number analyzed (Participants) | 8 | 7
score on a scale | 27 (14.1) | 24.7 (8.4)

2. Secondary Outcome: Patient Health Questionnaire
Description: The Patient Health Questionnaire (PHQ-9) is a reliable and valid 9-item measure of depression severity used to screen, diagnose, monitor, and measure the severity of depression. Scores can range from 0-27 and higher scores indicate greater depression severity.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RECLAIM/Intervention | Psychoeducation Materials Only/Control Group
Number analyzed (Participants) | 8 | 7
score on a scale | 6.4 (3.5) | 7.3 (4.2)

3. Secondary Outcome: Generalized Anxiety Disorder Scale
Description: The Generalized Anxiety Disorder Scale (GAD-7) is a brief 7-item measure for assessing generalized anxiety disorder. It consists of 7 questions and has a total score range from 0-21 and higher scores indicate greater frequency of anxiety symptoms.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RECLAIM/Intervention | Psychoeducation Materials Only/Control Group
Number analyzed (Participants) | 8 | 7
score on a scale | 10.4 (5.6) | 7.6 (4.4)

4. Secondary Outcome: Pain, Enjoyment, General Activity
Description: The Pain, Enjoyment, and General Activity (PEG) scale is a three-item assessment tool used to monitor chronic pain over time. Each item uses a numerical rating scale from 0 to 10. The scores on each of the 3 items (pain levels on average, pain interference with enjoyment, and pain interference with general activity) are summed and averaged to provide a score that will range from 0-10. Lower scores indicate minimal pain impact.
Time Frame: 1 Week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RECLAIM/Intervention | Psychoeducation Materials Only/Control Group
Number analyzed (Participants) | 8 | 7
score on a scale | 4.8 (3.2) | 4.5 (2.2)

5. Secondary Outcome: Five Facet Mindfulness Questionnaire
Description: The Five Facet Mindfulness Questionnaire (FFMQ-15) is a self-report scale that measures an individual's dispositional mindfulness across 5 distinct facets. Responses are made on a 5-point Likert scale, are totaled, and higher scores indicate greater mindfulness. The minimum possible score for each of the mindfulness facets is 3 and the maximum possible score is 15.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RECLAIM/Intervention | Psychoeducation Materials Only/Control Group
Number analyzed (Participants) | 8 | 7
score on a scale
  Mindfulness Facet: Observing | 12 (2.8) | 10 (1.4)
  Mindfulness Facet: Describing | 9.8 (3.4) | 10.4 (1.3)
  Mindfulness Facet: Awareness | 10.8 (2.9) | 10 (1.9)
  Mindfulness Facet: Non-judging | 11.3 (2.6) | 11.7 (2)
  Mindfulness Facet: Non-reacting | 10.1 (1.7) | 9.6 (1.3)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from enrollment until follow-up assessments were completed, which was approximately 4 months for all participants
Arm/Group | RECLAIM/Intervention | Psychoeducation Materials Only/Control Group
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

LIMITATIONS AND CAVEATS:
The investigators only included Veterans who were receiving VA care within one region of the country.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-30): https://cdn.clinicaltrials.gov/large-docs/08/NCT05975008/Prot_SAP_001.pdf
  • Informed Consent Form (2023-01-30): https://cdn.clinicaltrials.gov/large-docs/08/NCT05975008/ICF_000.pdf